CLINICAL TRIAL: NCT01647165
Title: Phase II Study of Subcutaneous (SC) Bortezomib, Lenalidomide and Dexamethasone for Relapsed and/or Refractory Multiple Myeloma; Followed by SC Bortezomib Maintenance
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120169; 12-C-0169
Record Dates: First submitted 2012-07-19; First posted 2012-07-20 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-03-11

CONDITIONS: Multiple Myeloma
Keywords: Maintenance Strategy; Plasma Cell Neoplasm; Proteasome Inhibitor; Immunomodulatory Drugs; Novel Therapy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Lenalidomide; Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Cycle 1-8: 1.0 mg/m2 SC at a concentration of 2.5 mg/ml or 1 mg/ml to the thighs or abdomen on days 1, 4, 8, 11 of a 21 day cycle for 8 cycles.
Drug: Lenalidomide — Cycle 1: 15 mg oral daily on days 2-14 of 21 day cycle; Cycle 2-8: 15 mg oral daily on days 1-14 of a 21 day cycle
Drug: Dexamethasone — Cycle 1: 10 mg oral or IV daily on days 2,4,5,8,9,11,12 of a 21 day cycle; Cycle 2-8: 10 mg oral or IV on days 1, 2, 4, 5, 8, 9, 11, 12 of a 21 day cycle

SUMMARY:
Background: Bortezomib is a drug approved by the Food and Drug Administration (FDA) to treat patients with multiple myeloma. It is given by intravenous injection. Lenalidomide is a drug that alters the immune system. It may also help suppress tumor growth. It is approved by the FDA to treat some types of blood cancers. Dexamethasone prevents or treats inflammation. It is sometimes used to treat multiple myeloma.

Objectives: The purpose of this study examine how the combination of the study drugs affects myeloma.

-

Eligibility:

* Participants at least 18 years old who have multiple myeloma that has come back, did not respond to treatment, or worsened while being treated.
* Participants who may be pregnant will be tested to ensure that they are not pregnant.

Design:

* Participants will be screened with a history and physical examination. Blood work and urine samples will be taken. A series of x-rays of all bones will be done. A bone marrow biopsy will be done.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Treatment will continue as long as the cancer does not grow or spread and no serious side effects develop.
* There will be up to eight 21-day treatment cycles.
* Bortezomib is given by subcutaneous (under the skin) (SC) injection on days 1, 4, 8, and 11 of the cycle.
* Lenalidomide is given by mouth on days 1 14 of the cycle.
* Dexamethasone is given by mouth on days 1, 2, 4, 5, 8, 9, 11, and 12 of the cycle.
* Following cycle eight, if the disease is stable or better, participants will receive bortezomib SC at the dose given at the end of cycle eight.
* Participants will take valacyclovir or acyclovir while taking bortezomib to prevent virus infections.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is an incurable plasma cell neoplasm with a median survival of 3-4 years.
* Increased survival has been achieved with the introduction of the proteasome inhibitor bortezomib and immunomodulatory drugs (IMiDs) such as lenalidomide. Bortezomib and lenalidomide have different but overlapping mechanism of anti-MM activity in preclinical studies.
* Despite the benefits of novel agents, bortezomib and lenalidomide pose clinical challenges. Bortezomib drug toxicity includes neuropathy, GI distress, myelosuppression and herpes zoster reactivation. Together with lenalidomide, the incidence of sensory neuropathy reaches 80%.
* Subcutaneous (SC) Bortezomib was evaluated in a prospective phase I trial for relapsed and/or refractory MM. SC administration was found to be comparable with the established IV route, with no differences in overall systemic availability and pharmacodynamic activity, similar toxicity profiles, and similar response rates.
* Combining SC, rather than IV bortezomib, with lenalidomide and dexamethasone is especially attractive given the potential for less overall neurotoxicity and improved convenience for the patient.
* Also, using bortezomib SC as a maintenance therapy after combination therapy is a novel strategy that has the potential to set the stage for coming oral proteasome inhibitors as potential maintenance strategies in the future.

Objectives:

Primary Objective

* Determine response rates, of S.C. bortezomib, lenalidomide, and dexamethasone (VRd) in relapse and/or refractory MM patients

Secondary Objectives

* Assess peripheral blood for immune cell populations in relation to SC bortezomib maintenance
* Evaluate toxicity, including peripheral neuropathy
* Evaluate patterns of change in patient-reported quality of life and symptom distress
* Gauge the feasibility, responsiveness to change and associated effect sizes when using patient-reported outcomes to augment clinician ratings of regimen-related treatment toxicity, including incidence and severity of peripheral neuropathy
* Determine duration of response
* Determine progression free survival

Eligibility:

* Patients with histologically confirmed relapsed and/or refractory multiple myeloma
* Age greater than or equal to 18 years
* Without serious co-morbidity that would interfere with receipt of VRd
* If patient has neuropathy, it must be less than or equal to Grade 1 at the time of first dose or within 14 days of enrollment
* Absolute neutrophil count (ANC) greater than equal to 1.0 K/uL, hemoglobin less than or equal to 8 g/dL, and platelet count greater than or equal to 75 K/uL
* Adequate hepatic function, with bilirubin < 1.5 times ULN; AST and ALT < 3.0 times ULN
* Creatinine Clearance greater than or equal to 60 ml/min. CrCl will be calculated by Cockcroft-Gault method. CrCl (calculated) = (140 Age) times Mass (in kilograms) times [0.85 if Female] 72 times Serum Creatinine (in mg/dL). If calculated CrCl based on Cockcroft-Gault method is < 60 mL/min, patient will have a 24 hr urine collection to measure CrCl. The measured CrCl must also be greater than or equal to 60 ml/min for the patient to be eligible.

Design:

Patient will receive treatment in this single arm study for 8 total cycles (each cycle is 21 days) with the following drugs, dosages and schedule:

- Bortezomib

Cycle 1-8: 1.0 mg/m(2) SC at a concentration of 2.5 mg/ml to the thighs or abdomen on days 1, 4, 8, 11 of 21 day cycle

- Lenalidomide

Cycle 1: 15 mg oral daily on days 2-14 of 21 day cycle

Cycle 2-8: 15 mg oral daily on days 1-14 of 21 day cycle

- Dexamethasone

Cycle 1: 10 mg oral on days 2,4,5,8,9,11,12 of 21 day cycle

Cycle 2-8: 10 mg oral on days 1,2,4,5,8,9,11,12 of 21 day cycle

- Maintenance therapy

After completion of cycle 8, patients with greater than or equal to stable disease will receive maintenance with bortezomib S.C. at a dose per end of Cycle 8. Maintenance will be given on days 1 and 15 of a 28 day cycle, and will continue until progression or unacceptable toxicity.

ELIGIBILITY:
* INCLUSION CRITERIA:

2.1.1.1 Relapsed and/or refractory histologically confirmed multiple myeloma as defined by:

1. Relapse from complete response with reappearance of the serum or urinary paraprotein, more or equal than 5% bone marrow plasma cells, new lytic bone lesions and /or soft tissue plasmacytomas, an increase in size of residual bone lesions and /or development of hypercalcemia (corrected serum calcium >11.5 mg/dl) not attributable to another cause.
2. Progressive disease: when a complete response has not been achieved, include new or expanding bone lesions, hypercalcemia, and a >25% increase in serum monoclonal paraprotein concentration, 24-hour urinary light chain excretion, or plasma cells within the bone marrow.
3. Refractory disease: Unresponsiveness to current therapy or progressive disease within 60 days of prior treatment.

2.1.1.2 Measurable disease within the past 4 weeks defined by any one of the following:

1. Serum monoclonal protein greater than or equal to 1.0 g/dL
2. Urine monoclonal protein >200 mg/24 hour
3. Serum immunoglobulin free light chain > 10 mg/dL AND abnormal

kappa/lambda ratio (reference 0.26-1.65)

2.1.1.3 Creatinine Clearance greater than or equal to 60 ml/min. CrCl will be calculated by Cockcroft-Gault method. CrCl (calculated) = (140 Age) times Mass (in kilograms) times [0.85 if Female] 72 times Serum Creatinine (in mg/dL). If calculated CrCl based on Cockcroft-Gault method is < 60 mL/min, patient will have a 24 hr urine collection to measure CrCl. The measured CrCl must also be greater than or equal to 60 ml/min for the patient to be eligible.

2.1.1.4 Age > 18 years

2.1.1.5 Eastern Cooperative Oncology Group (ECOG) performance status 0-2

2.1.1.6 Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of VELCADE, or agree to completely abstain from heterosexual intercourse.

2.1.1.7 Absolute neutrophil count (ANC) greater than or requal to 1.0 K/uL, hemoglobin greater than or equal to 8 g/dL (transfusions are permissible), and platelet count greater than or equal to 75K/uL within 7 days before enrollment.

2.1.1.8 Adequate hepatic function, with bilirubin < 1.5 times ULN; AST and ALT < 3.0 times ULN

2.1.1.9 Patients must have completed prior treatments (except steroids) at least 30 days before enrollment.

2.1.1.10 Prior allogeneic stem cell transplant without evidence of graft versus host disease. (GVHD) will be eligible at the investigator s discretion.

2.1.1.11 Permitted concurrent systemic treatment for MM.

1. Treatment of hypercalcemia or spinal cord compression or aggressively progressing myeloma with corticosteroids is permitted.
2. Bisphosphonates are permitted.
3. Radiotherapy is permitted. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

   2.1.1.12 All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist .

   2.1.1.13 Females of childbearing potential (FCBP) (Cross) must have a negative serum beta-human chorionic gonadotropin (beta-hCG) or urine pregnancy test within 10 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

   2.1.1.14 Male subjects, even if surgically sterilized (ie, status prostatectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.

   2.1.1.15 Subjects must be able to give voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

   2.1.1.16 Known HIV infected patients meeting the following characteristics are eligible:
   * CD4 cell count greater than or equal to 334/mm(3)
   * Meeting either of the following:
   * Willing to suspend antiretroviral therapy for duration of protocol therapy or
   * On stable regimen of combination antiretroviral therapy that does not include either zidovudine or stavudine for at least 12 weeks and without evidence of toxicity

   EXCLUSION CRITERIA:

   2.1.2.1 Refractory to lenalidomide and/or bortezomib in the most recent line of therapy

   2.1.2.2 Prior allogeneic stem cell transplant if the patient has graft versus host disease (GVHD).

   2.1.2.3 Plasma cell leukemia

   2.1.2.4 Pregnant or lactating females. Confirmation that the subject is not pregnant must be established by a negative serum <=-human chorionic gonadotropin (beta hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women.

   2.1.2.5 Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.

   2.1.2.6 Uncontrolled hypertension or diabetes

   2.1.2.7 Active hepatitis B or C infection

   2.1.2.8 Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.

   2.1.2.9 Has refractory GI disease with refractory nausea/vomiting, inflammatory bowel disease, or bowel resection that would prevent absorption

   2.1.2.10 Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance of study requirements

   2.1.2.11 Significant neuropathy greater than or equal to Grade 1 with pain or Grade 2 at the time of first dose or within 14 days of enrollment.

   2.1.2.12 Contraindication to any concomitant medication, including antivirals, anticoagulation prophylaxis, tumor lysis prophylaxis, or hydration given prior to therapy

   2.1.2.13 Active infection requiring treatment within two weeks prior to first dose

   2.1.2.14 Major surgery within 1 month prior to enrollment

   2.1.2.15 Hypersensitivity to bortezomib, boron, mannitol or lenalidomide

   2.1.2.16 Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.

   2.1.2.17 Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07-11; Primary Completion 2015-06-26 (Estimated); Study Completion 2015-06-26 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 2 years

SECONDARY OUTCOMES:
Progression-free survival | 3 years
Duration of response | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carl O Landgren, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. N Engl J Med. 2004 Oct 28;351(18):1860-73. doi: 10.1056/NEJMra041875. No abstract available. PMID 15509819
- [Background] Richardson PG, Weller E, Lonial S, Jakubowiak AJ, Jagannath S, Raje NS, Avigan DE, Xie W, Ghobrial IM, Schlossman RL, Mazumder A, Munshi NC, Vesole DH, Joyce R, Kaufman JL, Doss D, Warren DL, Lunde LE, Kaster S, Delaney C, Hideshima T, Mitsiades CS, Knight R, Esseltine DL, Anderson KC. Lenalidomide, bortezomib, and dexamethasone combination therapy in patients with newly diagnosed multiple myeloma. Blood. 2010 Aug 5;116(5):679-86. doi: 10.1182/blood-2010-02-268862. Epub 2010 Apr 12. PMID 20385792
- [Background] San Miguel JF, Schlag R, Khuageva NK, Dimopoulos MA, Shpilberg O, Kropff M, Spicka I, Petrucci MT, Palumbo A, Samoilova OS, Dmoszynska A, Abdulkadyrov KM, Schots R, Jiang B, Mateos MV, Anderson KC, Esseltine DL, Liu K, Cakana A, van de Velde H, Richardson PG; VISTA Trial Investigators. Bortezomib plus melphalan and prednisone for initial treatment of multiple myeloma. N Engl J Med. 2008 Aug 28;359(9):906-17. doi: 10.1056/NEJMoa0801479. PMID 18753647